CLINICAL TRIAL: NCT03111446
Title: General Anesthesia Versus Spinal Anesthesia in Patients of HELLP Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Talaat Mostafa, Dr., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SpinalHELLP
Record Dates: First submitted 2017-03-27; First posted 2017-04-12 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2017-04

CONDITIONS: HELLP Syndrome
MeSH Terms: conditions — HELLP Syndrome | interventions — Anesthesia, Spinal; Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spinal Anesthesia (Active Comparator): Spinal anesthesia will be used to anesthetize patients in this group for caesarian section
  Interventions: Procedure: Spinal Anesthesia
- General Anesthesia (Active Comparator): Standardized General Anesthesia will be used to anesthetize patients in this group for caesarian section
  Interventions: Procedure: General Anesthesia

INTERVENTIONS:
Procedure: Spinal Anesthesia — Spinal needle 25G with Quincke's bevel will be used. It will be induced with a total of 10 mg of 0.5% hyperbaric bupivacaine and 20 mcg fentanyl (total volume 2.4 ml) at the L3-4 interspace. The parturient will be returned to the supine position with a left lateral tilt of 15° to facilitate left uterine displacement. The upper sensory block level will be checked 5 min after the spinal injection by assessing the loss of cold sensation from alcohol swabs, to ensure that a Th6 sensory block level has been achieved.
  Arms: Spinal Anesthesia
Procedure: General Anesthesia — Pre-oxygenation with oxygen 100% via a tight fitting mask rapid sequence technique. Induction is by thiopental (5 mg kg lean body weight) and succinylcholine1.5 mg kg body weight), cricoid pressure should be applied before consciousness is lost and kept in place until confirmation of tracheal intubation with capnography and the cuff of the tracheal tube is inflated. Auscultating the chest helps exclude endobronchial intubation. At this point, surgery may commence.
  Arms: General Anesthesia

SUMMARY:
Anesthesia for caesarian section in patients with HELLP syndrome is a challenge. Measures should be taken during caesarian delivery to guard against the maternal and fetal complications associated with HELLP syndrome.

DETAILED DESCRIPTION:
The choice of anesthesia for caesarian section in parturient with HELLP syndrome is a debate. The low platelet count, associated with HELLP syndrome, has often favored the choice of general anesthesia for the caesarian delivery of these parturient. However, general anesthesia in such cases; is not a risk-free approach. General anesthesia is associated with increased risk of difficult airways, stress response to intubation and aspiration. It is also thought to have an effect on the fetus with the potential placental transfer of inhalational anesthetics prior to delivery.

Regional anesthesia is widely regarded as a means of providing analgesia for cesarean section.it also avoids the above-mentioned risks associated with general anesthesia. Regional anesthesia for caesarian section in patients with HELLP syndrome has been used by some researchers in many centers with encouraging results.

The lowest platelet count at which one can safely administer neuraxial anesthesia for labour and delivery is controversial. Published studies are few and sample sizes small.

Criteria developed at the University of Mississippi, as of 2006: "For a patient to merit a diagnosis of HELLP syndrome, class 1 requires severe thrombocytopenia (platelets ≤50,000/μl), evidence of hepatic dysfunction (AST and/or ALT ≥70 IU/l), and evidence suggestive of hemolysis (total serum LDH ≥600 IU/l); class 2 requires similar criteria except thrombocytopenia is moderate (>50,000 to ≤100,000/μl); and class 3 includes patients with mild thrombocytopenia (platelets >100,000 but ≤150,000/μl), mild hepatic dysfunction (AST and/or ALT ≥40 IU/l), and hemolysis (total serum LDH ≥600 IU/L).

The researchers chose to investigate class 2 HELLP syndrome as class 3 proved to be safe with regional anesthesia while class 1 seemed to be high risk and un-ethical to do spinal anesthesia with very low platelets count with lack of any evidence to its safety.

ELIGIBILITY:
Inclusion Criteria:

Patients with class (II) (12) HELLP syndrome scheduled for elective caesarian section:

Diagnosis of HELLP syndrome was based on the clinical diagnosis of preeclampsia and the following laboratory abnormalities (13):

1. Hemolysis: characteristic peripheral blood smear, serum lactic dehydrogenase (LDH) ≥ 600 U/ l, total bilirubin ≥ 1.2 mg /dl, decreased hemoglobin and hematocrit.
2. Elevated liver enzymes, defined as aspartate aminotransferase (AST). ≥ 70 U/ l, alanin aminotransferase (ALT) ≥ 50 U/ l and lactate dehydrogenase (LDH) ≥ 600 U/ l.
3. Low platelet count: class 2 HELLP having a platelet nadir between > 50000 and 100000 mm-3.

Exclusion Criteria:

1. Emergency cases
2. Placenta praevia
3. Cardiovascular or cerebrovascular disease.
4. Morbid obesity with a BMI ≥40
5. Gestational age <36 or >41 weeks
6. Platelet counts less than 50000 mm-3; class 1 HELLP and class 3 HELLP having platelet count more than 100 000 mm-3

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Parturients with HELLP syndrome presented for elective caesarian section
Enrollment: 60 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
The incidence of perioperative mortality in both groups. | up to one week postoperative
  Maternal

SECONDARY OUTCOMES:
occurence bradycardia | up to 24 hours postoperative
  heart rate less than 50 beat/min
occurrence of tachycardia | up to 24 hours postoperative
  heart rate more than 120 beats/min
occurrence of hypotension | up to 24 hours postoperative
  mean arterial blood pressure < 40% of the baseline
occurrence of hypertension | up to 24 hours postoperative
  mean arterial blood pressure > 40% of the baseline
incidence of cerebral hemorrhage | up to one week postoperative
  detected by CT in patients with neurological deficits

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided